CLINICAL TRIAL: NCT03908489
Title: Evaluation of Post-operative Pain After Vital Pulpotomy of Primary Molars Using Allium Sativum Oil Versus Mineral Trioxide Aggregate (MTA) : (A Pilot Study)
Brief Title: Evaluation of Post-operative Pain After Vital Pulpotomy in Primary Molars Using Allium Sativum Oil Versus MTA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Oma Ahmed Elgebaly, Assistnat lecturer in Pediatric Dentistry and Public Health Department Nahda University, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1441989
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Deep Caries

STUDY DESIGN:
Intervention Model Description: same patient will one molar indicated for vital pulpotomy on one side and on contralateral side
Who Masked: Investigator, Outcomes Assessor
Masking Description: The statistician, clinical and radiographic outcomes assessors will be blinded in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention we want to test vital pulpotomy using garlic oil (Experimental): interventional group as garlic oil pulpotomy dressed in zinc oxide powder
  Interventions: Procedure: vital pulpotomy primary molars using garlic oil
- control or comparator as mta vital pulpotomy in primary molars (Active Comparator): mta vital pulpotomy in primary molars
  Interventions: Procedure: vital pulpotomy using mta

INTERVENTIONS:
Procedure: vital pulpotomy primary molars using garlic oil — vital pulpotomy using garlic oil
  Other Names: vital pulpotomy primary molars using Allium sativium oil
  Arms: intervention we want to test vital pulpotomy using garlic oil
Procedure: vital pulpotomy using mta — mta vital pulpotomy
  Other Names: mta vital pulpotomy
  Arms: control or comparator as mta vital pulpotomy in primary molars

SUMMARY:
Preservation of the remaining vital portion of curiously exposed pulpal tissue in primary teeth, was one of the most frequent problems in pediatric dentistry. To solve this problem, pulpotomy therapy was introduced. Pulpotomy involves amputation of the coronal portion of affected or infected dental pulp, treatment of the remaining vital radicular pulp tissue surface should preserve the vitality and function of all or part of the remaining radicular portion of the pulp. Furthermore, it is an accepted procedure for treating both primary and permanent teeth with carious pulp exposures, several materials have been using for capping the radicular pulp after pulpotomy, these included formocresol, glutaraldehyde, ferric sulfate, and mineral trioxide aggregate.

Allium sativum is one of the most extensively researched medical plants and its antibacterial activity depends on allicin produced by the enzymatic activity of allinase (a cysteine sulfoxide lyase). Allicin and other thiosulfinates are believed to be responsible for the range of therapeutic effects reported for garlic. Garlic extract has been reported to inhibit growth of various gram-positive and gram-negative bacteria. Previous studies showed that A. sativum oil is used as new pulp medications and it offers a good healing potential, leaving the remaining pulp tissue healthy and functioning. MTA is a unique material with various advantages. It has been used successfully by pediatric dentists in a variety of clinical applications. However, its drawbacks especially its high cost, discoloration potential, difficulty in handling, and long setting time.

DETAILED DESCRIPTION:
1. Hypothesis This research adopts null hypothesis; it assumes that the use of the both garlic oil dressed in zinc oxide powder and MTA as vital pulpotomy dressing material have the same effects.
2. Trial design:

   Pilot study, two arms split mouth design with 1:1 allocation ratio. Patient's, clinical and radiographic outcomes assessors and statistician will be blinded in this study.
3. Methods

   Intervention

   A. Diagnostic procedure:

   • Clinical examination will be done on the dental clinic using mirror and probe.

   • Diagnosis of the cases will be performed according to guidelines of AAPD 2017 for treatment of vital pulp therapy in primary teeth.

   • Preoperative photographs will be taken
   * An individual XCP (Extension Cone Paralleling) index will be prepared for each patient by registering the bite to allow consistent comparisons of the radiographs.
   * Preoperative periapical radiograph will be taken.

   B. Intra operative procedure:

   • After randomly selecting which side will be in an intervention or control groups.

   • Apply topical anaesthesia.

   • Local anesthesia administration.

   • Rubber dam application and access cavity preparation will be established using a sterile bur.

   • Coronal pulp tissue will be removed using sharp large spoon excavator.

   • Apply wet cotton pellet for few minutes.

   • Then one side will be treated with Allium sativum oil dressed with zinc oxide powder -A. sativum oil paste, contralateral with MTA.

   • Then, a layer of zinc phosphate base will be placed over the dressing materials.

   • After that, those molars will be restored with stainless steel crowns and cemented using glass ionomer cement (GIC).

   C. Follow up:

   Follow up will be performed at 3, 6 and 9 months according to guidelines for clinical and radiographic evaluation.

   D. Criteria for discontinuing or modifying intervention:

   In case of unsuccessful outcomes of the intervention technique, the case will be managed by MTA pulpectomy.

   E. Strategies to improve adherence to intervention:

   • Face to face sessions with the patients to stress on the importance of follow up.

   • Oral hygiene measures.

   F. Concomitant care Oral hygiene measures.
4. Outcomes

<!-- -->

1. ry outcome 1. Post-operative Pain: Spontaneous pain and pain on biting will be reported by asking the patient using visual analogue scale
2. ry outcomes :

<!-- -->

1. Pain on percussion:Presence or absence of pain will be detected by tapping on the tooth using back of mirror handle using visual analogue scale.
2. Swelling:

   Presence or absence of swelling related to the affected tooth will be detected by visual intra-oral clinical examination.
3. Sinus or fistula:Presence or absence of sinus or fistula related to the affected tooth will be detected by visual intra-oral clinical examination.
4. Furcation involvement:It will be evaluated radiographically using DIGORA software using radiographic failure score.
5. periapical radiolucency: It will be evaluated radiographically using DIGORA software.
6. Pathological internal or external root resorption: It will be evaluated radiographically using DIGORA software.
7. Widening of periodontal membrane space:It will be evaluated radiographically using DIGORA software.

5- Recruitment: Recruitment of the patients will be from the outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Cairo University. Screening of patients will continue until the target population is achieved.

6- Implementation Co-supervisor; Randa Youssef Abd Al Gawad will assign which participant tooth will be included to either control or intervention groups according to the generated random sequence.

7. Masking/blinding: The statistician, clinical and radiographic outcomes assessors will be blinded in this study.

8. Data collection, management, and analysis: Data collection method

Baseline data will be collected by the operator through a paper-based Case Report custom made form (CRF) which will be developed by the research team. It will include the following items:

1. Patient serial number.
2. Demographic data.
3. Patients medical history:

   * Past medical history.
   * Any present disease or illness.
   * Current medication.
   * Any specific pre-treatment medication.
4. Past dental history.
5. Records for current dental condition (intra-oral examination and caries index).

The custom made CRF will be developed before online registration of the study protocol. CRF will be anonymous where patients will be identified by their serial number. The full detailed personal data of the patient will be written in a separate sheet having the patient's serial number for further contact with patient, this sheet can be only seen by the operator and the supervisors. The Co-supervisor; Dr. Randa Youssef Abd El-Gawad, will have the role to monitor the process of data collection and check if there is any incomplete CRF.

Primary and secondary outcomes will be collected by the lead researcher as follow:

1. Pain (spontaneous or on biting):

   Will be recorded by asking patient using visual analogue scale
2. Pain on percussion:

   Presence or absence will be detected by tapping the tooth with the back of the mirror using visual analogue scale
3. Swelling:

   Presence or absence will be detected by visual examination.
4. Sinus or fistula:

   Presence or absence will be detected by visual examination.
5. Widening in periodontal membrane space
6. furcation involvement or periapical radiolucency :Presence or absence will be detected radiographically by Digora Image plate according to radiographic failure score.

9- Data management: Data will be entered on a software then stored online on a Google app (Google drive). Only the lead researcher will be allowed to enter the data and it will be revised by both senior and co supervisors. Patient files will be stored in numerical order and stored in secure and accessible place and all data will be maintained in storage for 1 year after completion of the study.

Plans to promote participant retention and complete follow- up:

Telephone numbers of all patients included in the study will be recorded as a part of the written consent. All patients will be given a phone call at the time of the pre-determined follow up dates.

10 - Data monitoring: Monitoring No formal data monitoring committee will be needed since most of studies in Faculty of Dentistry are with known minimal risks.

11- Harms Any possible adverse effects of the interventions (allergy to any of the used materials, swelling, sinus, fistula, pain or infection) will be recorded.

12- Audit

Procedures for auditing include:

* Participant enrolment.
* Consent.
* Eligibility criteria.
* Allocation to study groups.
* Adherence to trial interventions.
* Outcomes assessment.

Auditing will be performed in order to preserve the integrity of the trial. This will be ensured by periodic independent review of trial processes and documents by the Evidence Based Committee, Faculty of Dentistry, Cairo University IV. Ethics and dissemination

13- Research ethics approval This protocol and the template informed consent forms appended to the protocol will be reviewed by the Ethics Committee of Scientific Research, Faculty of Dentistry, Cairo University.

14- Protocol amendments The Ethics Committee and Evidence Based Committee, Faculty of Dentistry, Cairo University will be notified of any administrative changes or modifications of the protocol which may impact on the conduct of the study, potential benefit of the patient or may affect patient safety, including changes of study objectives, study design, sample sizes or study procedure.

15- Informed consent Once the child is identified as eligible to the study by the clinical investigator, the trial procedures, benefits from the study and expected harms will be clearly discussed with parent or the child's legal guardian. This explanation will be simplified with avoidance of any pain promoting words when the trial is discussed with the child. Verbal assent will be obtained orally from the eligible child and the written consent will be signed by the child's guardians.

16- Confidentiality Personal information about participants will be acquired during the process of trial recruitment, eligibility screening, and data collection. Most of this information consists of private details. All study-related information will be stored securely at the study site. All participants' information will be stored in locked file cabinets in areas with limited access. All records that contain names or other personal identifiers, will be stored separately from study records identified by code number. All reports, data collection, process, and administrative forms will be identified by the child's ID (ticket serial number) and will not contain any personal information to protect the participant's confidentiality.

17- Declaration of interest No known conflict of interests.

18- Access to data Lead researcher, Nourhan Omar Elgebaly, will be given an access to the data sets. All data sets will be password protected. To ensure confidentiality, data dispersed to project team members will be blinded of any identifying participant information.

19- Ancillary and Post-trial care

• Final restoration of the teeth participated at the trial will be done in the same visit.

• All patients will be followed up until 9 months.

• Full mouth treatment in addition to preventive measures will be offered for all participants.

• Patients will be instructed to follow up the teeth one year after the end of the trial.

20- Dissemination policy

* Study results will be published as partial fulfillment of the requirements for PHD degree in Pediatric Dentistry.
* The result of the trial are intended to be disseminated in the library of the Faculty and in the Egyptian Dental Journal.
* Topics suggested for presentation or publication will be circulated to the authors.
* If results show the advantage of one intervention over the other, it will be recommended to be performed as a routine procedure during dental treatment.
* Thesis defence after completion of the study will be done in public with external judges.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy cooperative children with pair of contralateral deep carious mandibular primary molars indicated for vital pulpotomy.
2. In age range from 4 to 8 years.
3. Both sexes are included.
4. Patients with provoked pain.
5. Remaining radicular tissue is vital without suppuration or purulence.
6. With no clinical or radiographic signs of pulp necrosis.
7. Restorable teeth

Exclusion Criteria:

1. Excessive haemorrhage that cannot stop by a damp cotton pellet after several minutes
2. With congenital anomalies in teeth e.g., taurodontism, concrescence or fusion. 3- Patients who will show allergic reaction to any material will be used in this trial.

4- Will not be able to stick to follow up protocol in the trial and refuse to give communication data.

5- Patient's guardians refuse to sign up an informed consent before participating in this trial.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
post- operative Pain ( Spontaneous or on biting): | 3 months
  Pain ( Spontaneous or on biting) using visual analogue scale range from (0 -10) (0) No pain (10) the worst pain condition
post-operative pain (spontaneous or on bitting): visual analogue scale | at 6 months
  pain (spontaneous or on bitting) using visual analouge scale range from (0 -10) (0) No pain (10) the worst pain condition
post- operative Pain ( Spontaneous or on biting): visual analogue scale | at 9 months
  pain (spontaneous or on bitting) using visual analogue scale. range from (0 -10) (0) No pain (10) the worst pain condition

SECONDARY OUTCOMES:
periapical radiolucency | 3 months
  periapical radiolucency Binary (+/-)
  DIGORA ® for windows software.
periapical radiolucency | 6 months
  periapical radiolucency Binary (+/-)
  DIGORA ® for windows software.
periapical radiolucency | at 9 months
  periapical radiolucency Binary (+/-)
  DIGORA ® for windows software.
Pathologic internal or external root resorption | 3 months
  DIGORA ® for windows software. Binary (+/-)
Pathologic internal or external root resorption | 6 months
  DIGORA ® for windows software. Binary (+/-)
Pathologic internal or external root resorption | 9 months
  DIGORA ® for windows software. Binary (+/-)
Furcation involvement | 3 months
  DIGORA ® for windows software using furcation failure scores
Furcation involvement | 6 months
  DIGORA ® for windows software using furcation failure scores
Furcation involvement | 9 months
  DIGORA ® for windows software using furcation failure scores
Widening in the periodontal membrane space. DIGORA ® for windows software. Binary (+/-) | 3 months
  DIGORA ® for windows software. Binary (+/-)
Widening in the periodontal membrane space. DIGORA ® for windows software. Binary (+/-) | 6 months
  DIGORA ® for windows software. Binary (+/-)
Widening in the periodontal membrane space. DIGORA ® for windows software. Binary (+/-) | 9 months
  DIGORA ® for windows software. Binary (+/-)
Pain on percussion Back of the mirror: visual analogue scale | 3 months
  Back of the mirror (using visual analogue scale) range from (0 -10) (0) No pain (10) the worst pain condition
Pain on percussion Back of the mirror: visual analogue scale | 6 months
  Back of the mirror (visual analogue scale) range from (0 -10) (0) No pain (10) the worst pain condition
Pain on percussion Back of the mirror: visual analogue scale | 9 months
  Back of the mirror. (visual analogue scale) range from (0 -10) (0) No pain (10) the worst pain condition
Swelling Clinical examination by operator. Binary (+/-) | 3 months
  Clinical examination by operator. Binary (+/-)
Swelling Clinical examination by operator. Binary (+/-) | 6 months
  Clinical examination by operator. Binary (+/-)
Swelling Clinical examination by operator. Binary (+/-) | 9 months
  Clinical examination by operator. Binary (+/-)
Sinus or fistula Clinical examination by operator. Binary (+/-) | 3 months
  Clinical examination by operator. Binary (+/-)
Sinus or fistula Clinical examination by operator. Binary (+/-) | 6 months
  Clinical examination by operator. Binary (+/-)
Sinus or fistula Clinical examination by operator. Binary (+/-) | 9 months
  Clinical examination by operator. Binary (+/-)

CONTACTS AND LOCATIONS:
Overall Officials: cairo university, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
after thesis defense. the study will be published internationally to be available for everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one and half year.
Access Criteria: not yet